## Effects of Argan Spinosa Oil in the Treatment of Diaper Dermatitis in Infants and Toddlers: A Quasi-Experimental Trial

## **Informed Consent**

**Study Date:** 

1- February- 2018 Till 1-June-2019

## Approval to participate in scientific research

You are invited to participate in a scientific research that will be conducted by researchers from Jordan University of Science and Technology. We ask that you read the information carefully and calmly. You can also ask for clarifications or additional information about anything mentioned in this form or about this research as a whole from the main researcher.

**Research title:** Effects of Argan Spinosa Oil in the Treatment of Diaper Dermatitis in Infants and Toddlers: A Quasi-Experimental Trial.

<u>The main researchers:</u> Dr. The Nihaeih Al-Shayyab and Eman Al-Satari <u>Address:</u> Jordan University of Science and Technology - College of Nursing

**Phone:** 000962799373908

Research Objectives: to measure the effectiveness of the traditional medicinal product of Argan Spinosa Oil on the speed up of the healing process and alleviation of the symptoms with that of topical hydrocortisone 1% ointment on cases of dipper dermatitis in children aged two years or younger at the enrollment day, third day and at the seventh days of the end of the treatment. Furthermore, this study aimed to investigate variables that might increase the development of diaper dermatitis among these children.

<u>What you need to do</u>: We will ask you to use the provided medical product by the pediatrician during the study period which is seven consecutive days, and visits by the researcher will be made on the third and seventh days to measure the effectiveness of the product.

<u>Negative effects of participation in this research:</u> It is not expected that there will be any negative effect from participation in this research.

**Benefits:** The expected results of a medical product provided by a pediatrician accelerate the healing process and reduce symptoms of dermatitis caused by wearing diapers in infants / young children who participating in the study.

<u>Confidentiality:</u> Researchers undertake not to disclose the results of the research or give it to you unless you agree to participate in this study, your name will remain confidential and no person will have the right to see your medical or personal information.

<u>Participant approval:</u> I have clearly seen the content of the aforementioned scientific research. The researchers undertake not to disclose the results of the research or give it except to the person concerned. Accordingly, I voluntarily agree to participate in this research, and I know that the researchers will be ready to answer any questions. I know that I can revoke consent at any time, even if after signing, and a copy of this form the researchers will be given.

| Participant Signature | Participant Name |
|-----------------------|------------------|
| Researchers Signature | Date and Time |